CLINICAL TRIAL: NCT06918964
Title: Efficacy and Safety of Transcutaneous Auricular Vagus Nerve Stimulation for Acute Intracerebral Hemorrhage
Brief Title: TaVNS for Acute Intracerebral Hemorrhage
Acronym: TAVANS-ICH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Kaijiang Kang, Principal Investigator, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KangKJ
Record Dates: First submitted 2025-03-06; First posted 2025-04-09 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral Hemorrhage; taVNS; perihemtomal edema; neuroinflammation; secondary brain injury
MeSH Terms: conditions — Cerebral Hemorrhage; Neuroinflammatory Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and outcome assessors are unaware of the trial grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- taVNS intervention (Active Comparator): Patients will receive taVNS therapy twice daily for 10 consecutive days, in addition to receiving guideline-adherent conventional treatment during hospitalization.
  Interventions: Device: transcutaneous auricular vagus nerve stimulation device
- Sham taVNS intervention (Sham Comparator): Patients will receive sham taVNS twice daily for 10 consecutive days, in addition to receiving guideline-adherent conventional treatment during their hospital stay.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation device — Place the stimulation device on the left auricle and set the stimulation parameters according to the following conditions: a. Waveform: biphase, square wave; b. Wave width: 200 μs; c. Frequency: Alternating between low frequency (4 Hz for 4 s), high frequency (40 Hz for 8 s), and a 4 s pause; d. Intensity: The maximum intensity that induces the strongest sensation the individual can tolerate without causing pain, usually 1.5-3.5 mA; e. Treatment duration: Each treatment lasted 30 minutes, twice daily (8:00, 16:00) for 10 days.
  Arms: taVNS intervention
Device: Sham device — The sham taVNS group received the same parameters with a current intensity of 0.06 mA.
  Arms: Sham taVNS intervention

SUMMARY:
This study aims to evaluate the efficacy and safety of transcutaneous auricular vagus nerve stimulation (taVNS) in patients with acute intracerebral hemorrhage (ICH). The taVNS intervention will be delivered using the BS-TVNS800-1 transcutaneous electrical stimulation therapy device (KERFUN, Shanxi, China). A total of 186 patients will be randomly assigned in a 1:1 ratio to either the taVNS group or the sham-taVNS group. The primary outcome is the relative volume of perihematoma edema assessed on day 10-14 after randomization. Adverse events associated with taVNS therapy will be systematically evaluated to assess its safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with spontaneous supratentorial intracerebral hemorrhage.
2. Age between 18 and 80 years.
3. Onset within 72 hours.
4. Hematoma volume between 5 and 40 mL.
5. Glasgow Coma Scale (GCS) score greater than 8.
6. Written informed consent obtained from the patient or their legal representative.

Exclusion Criteria:

1. Secondary intracerebral hemorrhage (e.g., traumatic, tumor-related, vascular malformation, aneurysm, or coagulopathy-related).
2. Primary intraventricular hemorrhage.
3. Parenchymal hemorrhage that ruptures into the ventricles, with blood completely filling one lateral ventricle, the third ventricle, the fourth ventricle or more than half of both lateral ventricles.
4. Progressive neurological or other severe diseases.
5. Planned surgical treatment within 24 hours.
6. Pre-existing disability caused by previous illnesses: Modified Rankin Scale (mRS) score ≥ 3.
7. Patients with severe cardiomyopathy, heart failure, pacemaker implantation, atrial fibrillation, frequent premature beats, second-degree or higher atrioventricular block, or other severe arrhythmias.
8. Severe pulmonary disease, liver disease, renal insufficiency (glomerular filtration rate < 30 mL/min), active gastrointestinal bleeding, or malignant tumors with an expected survival of less than 3 months.
9. Patients with hyperthyroidism, hypothyroidism, syncope, epilepsy, multiple sclerosis, Parkinson's disease, multiple system atrophy, or other known disorders affecting autonomic nervous function.
10. Use of medications that interfere with autonomic function (e.g., beta-blockers, theophylline, tricyclic antidepressants, or steroids) within 7 days before screening.
11. Patients who cannot tolerate taVNS.
12. Congenital or acquired ear abnormalities preventing taVNS treatment.
13. Inability to comply with 10 days of treatment.
14. Pregnancy or within 30 days of delivery.
15. Participation in another interventional clinical trial.
16. Inability to obtain written informed consent from the participant or their legal representative.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Volume of perihematoma edema assessed by CT | Day 10-14 after randomization
  Relative edema volume.

SECONDARY OUTCOMES:
Autonomic activity assessed by heart rate variability | Day 10-14 after randomization
  Heart rate variability (HRV) will be assessed using a 10-minute electrocardiogram (ECG) recorded with a 12-lead ECG Holter (TeleECG BI 12E, Biomedical Instruments Co., Ltd., Shenzhen). HRV indices will be analyzed in both the time domain (e.g., SDNN, RMSSD) and the frequency domain (e.g., LF, HF, LF/HF).
Autonomic activity assessed by baroreflex sensitivity | Day 10-14 after randomization
  Baroreflex sensitivity (BRS) will be evaluated by noninvasively measuring beat-to-beat signals for 10 min using a servo-controlled plethysmograph (FMS-8A, Delica Medical Equipment Co., Ltd., Shenzhen) placed on the middle finger.
National Institutes of Health stroke scale (NIHSS) | Day 10-14 after randomization
  NIHSS is used to assess the severity of functional impairment caused by stroke. It consists of 11 test items, with a total score ranging from 0 to 42. A higher score indicates a more severe stroke.
GCS (Glasgow Coma Scale) | Day 10-14 after randomization
  The GCS is used to assess the level of consciousness in patients, with the total score ranging from 3 to 15. Lower scores indicate more severe impairment.
MMSE (Mini-Mental State Examination) | Day 10-14 after randomization
  The Mini-Mental State Examination (MMSE) is a widely used cognitive screening tool designed to assess global cognitive function, including orientation, memory, attention, language, and visuospatial skills. Scores range from 0 to 30, with higher scores indicating better cognitive performance.
MoCA (Montreal Cognitive Assessment) | Day 10-14 after randomization
  The Montreal Cognitive Assessment (MoCA) is another cognitive screening instrument optimized for detecting mild cognitive impairment (MCI) and early dementia. Scores range from 0 to 30, with higher scores indicating better cognitive performance.
PHQ-9 (Patient Health Questionnaire-9) | Day 10-14 after randomization
  The Patient Health Questionnaire-9 (PHQ-9) is a brief, self-report tool validated for screening and monitoring depression severity. Scores range from 0 to 27, with higher scores reflecting greater symptom severity.
90-day National Institutes of Health stroke scale (NIHSS) | 90 ± 7 days after randomization
  NIHSS is used to assess the severity of functional impairment caused by stroke. It consists of 11 test items, with a total score ranging from 0 to 42. A higher score indicates a more severe stroke.
90-day modified Rankin Scale (mRS) | 90 ± 7 days after randomization
  The mRS is used to measure the degree of disability or dependence after a stroke. The scale ranges from 0 to 6 and higher scores indicate greater functional impairment.
90-day EQ-5D (EuroQol 5-Dimension Questionnaire) score | 90 ± 7 days after randomization
  The EQ-5D is a standardized instrument used to assess health-related quality of life.
90-day GCS (Glasgow Coma Scale) | 90 ± 7 days after randomization
  The GCS is used to assess the level of consciousness in patients, with the total score ranging from 3 to 15. Lower scores indicate more severe impairment.
90-day MMSE (Mini-Mental State Examination) | 90 ± 7 days after randomization
  The Mini-Mental State Examination (MMSE) is a widely used cognitive screening tool designed to assess global cognitive function, including orientation, memory, attention, language, and visuospatial skills. Scores range from 0 to 30, with higher scores indicating better cognitive performance.
90-day MoCA (Montreal Cognitive Assessment) | 90 ± 7 days after randomization
  The Montreal Cognitive Assessment (MoCA) is another cognitive screening instrument optimized for detecting mild cognitive impairment (MCI) and early dementia. Scores range from 0 to 30, with higher scores indicating better cognitive performance.
90-day PHQ-9 (Patient Health Questionnaire-9) | 90 ± 7 days after randomization
  The Patient Health Questionnaire-9 (PHQ-9) is a brief, self-report tool validated for screening and monitoring depression severity. Scores range from 0 to 27, with higher scores reflecting greater symptom severity.

OTHER OUTCOMES:
Safety assessment | In the 10-day treatment period
  Adverse events, serious adverse events, death
Perihematomal blood-brain barrier permeability | Day 5-7 after randomization
  Perihematomal blood-brain barrier permeability will be assessed by Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI).
Evaluation of glymphatic system | Day 5-7 after randomization
  Impairment of the function of the glymphatic system will be assessed by diffusion kurtosis imaging analysis along the perivascular space (DKI-ALPS).
Assessment of microglial activation | Day 7-9 after randomization
  Microglial activation will be quantified by TSPO-PET/MRI.
Interleukin-1β (IL-1β) level in peripheral blood | Day 10-14 after randomization
  IL-1β: A pro-inflammatory cytokine (measured in pg/mL) that drives fever, neutrophil activation, and autoimmune responses. It will be detected by ELISA.
Interleukin-6 (IL-6) | Day 10-14 after randomization
  IL-6: A pro-inflammatory cytokine (pg/mL) involved in acute-phase protein synthesis and B-cell differentiation, and implicated in infections. It will be detected by ELISA.
Tumor Necrosis Factor-alpha (TNF-α) | Day 10-14 after randomization
  TNF-α is a pro-inflammatory cytokine (pg/mL) which can be detected via ELISA.
Interleukin-4 (IL-4) | Day 10-14 after randomization
  IL-4 is an anti-inflammatory Th2 cytokine (pg/mL) which will be measured by ELISA.
Interleukin-10 (IL-10) | Day 10-14 after randomization
  IL-10 is an anti-inflammatory regulator (pg/mL), which will be quantified via ELISA.
Transforming Growth Factor-beta (TGF-β) | Day 10-14 after randomization
  TGF-β is a multifunctional cytokine (pg/mL) that is involved in regulation of cell growth, differentiation, and apoptosis. It will be detected by ELISA.
Neurofilament light chain (NFL) | Day 10-14 after randomization
  NFL is a non-specific biological marker representing neuronal injury (measured in pg/mL). It will be measured by ELISA.
Monocyte subsets | Day 10-14 after randomization
  Classical (CD14++CD16-) differentiate into macrophages for tissue repair, non-classical (CD14+CD16++) patrol vasculature for surveillance, measured in cells/μL by flow cytometry.
CD4+ T cells | Day 10-14 after randomization
  Coordinate adaptive immunity (helper role, cells/μL) via cytokine secretion and immune activation, assessed by flow cytometry with surface marker staining.
CD8+ T cells | Day 10-14 after randomization
  Mediate cytotoxicity (cells/μL), quantified using flow cytometry.
NK cells | Day 10-14 after randomization
  Innate lymphocytes (cells/μL) detected via flow cytometry.
B cells | Day 10-14 after randomization
  Produce antibodies for humoral immunity (measured in cells/μL), enumerated by flow cytometry (CD19/CD20 markers).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes